CLINICAL TRIAL: NCT03154216
Title: The Effect of Milk as a Recovery Beverage After Exercise on Next-day Postprandial Triglycerides
Brief Title: Milk as a Recovery Beverage After Exercise for Improving Metabolic Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Collaborators: Dairy Farmers of Canada (Other)
Responsible Party: Principal Investigator, Phil Chilibeck, Professor, University of Saskatchewan
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 16-300
Record Dates: First submitted 2017-05-12; First posted 2017-05-16 (Actual); Last update posted 2019-05-07 (Actual); Status verified 2019-05

CONDITIONS: Hyperlipemia, Carbohydrate Inducible
MeSH Terms: conditions — Hyperlipoproteinemia Type IV | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise only (Experimental): 90 minutes of exercise
  Interventions: Behavioral: Exercise
- Exercise and high glycemic index drink (Experimental): 90 minutes of exercise followed by consumption of high-glycemic index Gatorade drink matched for calories expended during the exercise
  Interventions: Behavioral: Exercise; Other: Drink
- Exercise and low glycemic index drink (Experimental): 90 minutes of exercise followed by consumption of low-glycemic index milk drink matched for calories expended during the exercise
  Interventions: Behavioral: Exercise; Other: Drink
- No exercise and no beverage (No Intervention): No exercise and no beverage

INTERVENTIONS:
Behavioral: Exercise — 90 minutes of moderate-intensity walking exercise on a treadmill
  Arms: Exercise and high glycemic index drink; Exercise and low glycemic index drink; Exercise only
Other: Drink — Beverage to be consumed after exercise
  Arms: Exercise and high glycemic index drink; Exercise and low glycemic index drink

SUMMARY:
Fasting blood fat levels (triglycerides) are often used to assess risk of heart disease but the level of fats in the blood after a meal is actually a stronger risk factor. Most of our day is spent digesting the food we eat (which takes hours). Therefore, "after meal" blood fat levels have more of an impact on formation of blockages in our arteries and our risk of heart disease compared to "fasting" blood fat levels. Exercise performed hours before a meal reduces the level of fats that appear in the blood after a meal and can be used to reduce our risk of heart disease. Exercise has this effect because muscle burns fats for hours after an exercise session is over; this helps to remove fats from the blood. Unfortunately, when high-sugar drinks (such as Gatorade) are consumed after exercise, the possible benefits of exercise for reducing blood fat levels after meals is lessened. This is because high-sugar drinks stimulate the release of insulin into the blood. Insulin is a hormone which inhibits fat burning at the muscle. Previous research we did showed that foods that result in a slower rise in blood sugar and lower release of insulin preserve the beneficial effects of exercise for lowering blood fat levels after the next meal. Milk also results in a slow rise in blood sugar and low release of insulin; therefore, it may also have this beneficial effect if consumed as a recovery beverage after exercise. Our proposed research will test the effects of consuming two popular exercise-recovery drinks (Milk vs. Gatorade) on the rise in blood fat levels after a meal given hours later. A total of 20 obese or overweight participants will take part. We predict that milk consumed after an exercise session in the evening will result in a lower increase in insulin, a greater amount of fat-burning at muscle and a lower blood fat level after a meal given the next morning. Milk and Gatorade are both promoted as good beverages to promote recovery after exercise. This study will provide evidence about milk as a healthier choice compared to Gatorade and will allow dairy producers to promote health benefits of dairy products.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death in Canada with annual direct and indirect costs estimated at $22 billion. Fasting lipid levels are associated with elevated risk of cardiovascular disease; however, postprandial lipids - the level of TG after a meal, are very potent predictors of cardiovascular disease risk because most of an individual's day is spent in the postprandial state. This problem is especially evident in obese individuals, who have an elevated postprandial TG response. An acute session of exercise is beneficial for reducing postprandial TG; however, caloric consumption immediately after exercise can attenuate this beneficial effect.

Carbohydrate quality may influence postprandial lipid response. Carbohydrates can be classified by their glycemic index (GI), where high GI carbohydrates are rapidly digested and result in large elevations in blood glucose. Low GI carbohydrates are digested slowly and result in a smaller, more gradual rise in blood glucose. High GI carbohydrates are associated with an elevated risk of cardiovascular disease and increased weight gain; whereas low GI carbohydrates are associated with a reduced risk of cardiovascular disease and decreased weight gain. As mentioned above, one of the main benefits of an acute session of exercise is to reduce TG levels after a subsequent meal. For example, an evening exercise session reduces the blood TG response after a high-fat breakfast provided the next day. This effect is negated if high GI beverages (i.e. sugar-sweetened drinks) are consumed immediately after exercise. Sports drinks such as Gatorade, and skim milk or chocolate milk are the leading beverages promoted for consumption during recovery after exercise. Gatorade has a high GI (i.e. GI=89) due to the inclusion of high amounts of simple sugars, whereas milk has a low GI (i.e. GI=34). Milk may therefore be a healthier choice for consumption after exercise.

No study has determined the effects of consuming low GI milk after an exercise session on next-day postprandial TG. Considering that consuming beverages after exercise is common practice and can influence blood lipid profiles, investigation into effects of low GI milk versus high GI recovery beverages is required.

The aim of this proposal is to determine if replacing calories expended during an evening session of endurance exercise with low GI milk can improve postprandial TG after a meal the next morning. We propose to look at the effects of consuming skim milk compared to Gatorade after endurance exercise on the blood TG, other lipids, glucose levels, and blood pressure responses after a high-fat meal consumed the morning after the exercise.

Our objective is to determine the effect of consuming milk after an evening exercise session on blood triglyceride response to a high fat meal the next morning. This will be compared to: A condition where exercise is performed followed by consumption of a high glycemic index Gatorade beverage; a condition where only exercise is performed with no after-exercise caloric consumption; a condition where neither exercise nor beverage is consumed in the evening. After each of these conditions, a high fat breakfast will be consumed the following morning (about 10 hours after the end of the exercise session). Blood will be collected before the breakfast and for 6 hours after the breakfast to determine postprandial metabolic response.

Our secondary objectives are to determine the effect of each condition on postprandial insulin, high density lipoprotein, apolipoprotein B, total cholesterol, and free fatty acids, and muscle fat oxidation. Blood pressure will also be assessed immediately after the evening exercise session and beverage consumption and continue throughout the night and throughout the postprandial period the next day.

Our primary hypothesis is that consuming low glycemic index milk after the evening exercise session will be superior to consuming Gatorade for reducing postprandial triglycerides the next morning.

Our secondary hypotheses are that consuming low glycemic index milk after the evening exercise session will be superior to consuming Gatorade for improving other metabolic measures (i.e. increasing high density lipoproteins, plasma free fatty acids, and fat oxidation, and reducing apolipoprotein B, low density lipoproteins, total cholesterol, and blood pressure) during the postprandial period after a high-fat meal.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index of 25 or greater
* 18-44 years of age

Exclusion Criteria:

* diabetics
* smokers
* those taking medications for cholesterol or glucose
* those who are allergic to milk

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-20 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-01-01 (Actual)

PRIMARY OUTCOMES:
Change in blood triglycerides | Change from baseline to 6 hours
  Triglyceride levels after a high-fat breakfast

SECONDARY OUTCOMES:
Change in blood glucose | Change from baseline to 6 hours
  Glucose levels after a high-fat breakfast
Change in fat oxidation | Change from baseline to 6 hours
  Fat oxidation after a high-fat breakfast
Change in low density lipoproteins | Change from baseline to 6 hours
  Low density lipoproteins after a high-fat breakfast
Change in high density lipoproteins | Change from baseline to 6 hours
  High density lipoproteins after a high fat breakfast
Change in total cholesterol | Change from baseline to 6 hours
  Total cholesterol after a high-fat breakfast
Change in insulin level | Change from baseline to 6 hours
  Insulin level after a high-fat breakfast
Change in blood pressure | Change from baseline to 16 hours
  Blood pressure after exercise and beverage consumption

CONTACTS AND LOCATIONS:
Overall Officials: Philip Chilibeck, PhD, Principal Investigator — University of Saskatchewan
Locations (1):
- College of Kinesiology, University of Saskatchewan, Saskatoon, Saskatchewan (SK), Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kaviani M, Chilibeck PD, Yee P, Zello GA. The effect of consuming low- versus high-glycemic index meals after exercise on postprandial blood lipid response following a next-day high-fat meal. Nutr Diabetes. 2016 Jul 4;6(7):e216. doi: 10.1038/nutd.2016.26. PMID 27376698
- [Derived] Gao R, Rapin N, Elnajmi AM, Gordon J, Zello GA, Chilibeck PD. Skim milk as a recovery beverage after exercise is superior to a sports drink for reducing next-day postprandial blood glucose and increasing postprandial fat oxidation. Nutr Res. 2020 Oct;82:58-66. doi: 10.1016/j.nutres.2020.08.007. Epub 2020 Aug 19. PMID 32977252